CLINICAL TRIAL: NCT06983028
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Atacicept in Multiple Autoimmune Glomerular Diseases (PIONEER)
Brief Title: Atacicept in Multiple Glomerular Diseases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT-001-0060
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: pMN; IgAN; Nephrotic Syndrome; MCD; FSGS
Keywords: IGA Glomerulonephritis; IGA Nephropathy; Iga Nephropathy 1; Immunoglobulin A Nephropathy Nephritis; IGA Type Nephropathy, IGA; Primary Membranous Nephropathy; Nephrotic Syndrome; Immunoglobulin A (IgA); Immunoglobulin A vasculitis with nephritis (IgAVN); Anti-PLA2R associated membranous nephropathy (PLA2R-MN); Idiopathic/primary nephrotic syndrome (MCD/FSGS); Urologic Diseases; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Male Urogenital Diseases; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases; Kidney Diseases; Glomerulonephritis, IGA
MeSH Terms: conditions — Nephrotic Syndrome; Macular dystrophy, corneal type 1; Glomerulonephritis, IGA; Urologic Diseases; Female Urogenital Diseases; Female Urogenital Diseases and Pregnancy Complications; Urogenital Diseases; Male Urogenital Diseases; Glomerulonephritis; Nephritis; Autoimmune Diseases; Immune System Diseases; Kidney Diseases | interventions — TACI receptor-IgG Fc fragment fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IgAN or IgAVN (Experimental): Adult and pediatric patients with biopsy proven IgAN or IgAVN with varied severity of proteinuria and kidney function beyond what is currently included in most clinical trials. Adults with post-transplant IgAN recurrence are also included.
  Interventions: Drug: Atacicept
- pMN (Experimental): Adults with biopsy-proven pMN associated with anti-PLA2R antibodies at low risk of spontaneous remission, or experiencing recurrent or resistant disease.
  Interventions: Drug: Atacicept
- Primary Nephrotic Syndrome (MCD/FSGS) (Experimental): Adults with biopsy-proven primary MCD or FSGS and evidence of anti-nephrin antibodies. Children with frequently relapsing, steroid-dependent, or non-genetic steroid-resistant nephrotic syndrome with evidence of anti-nephrin antibodies.
  Interventions: Drug: Atacicept

INTERVENTIONS:
Drug: Atacicept — Atacicept 150 mg SC QW via pre-filled syringe

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of atacicept in adult and adolescent participants and to measure the effect in reducing proteinuria and preserving renal function.

DETAILED DESCRIPTION:
The study will assess the safety and efficacy of atacicept in multiple autoimmune glomerular diseases including IgAN (IgA Nephropathy), pMN (Primary Membranous Nephropathy) and MCD/FSGS (Minimal Change Disease/Focal Segmental Glomerulosclerosis) in participants ages 10 and above with weekly SC injections.

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 40 kg
* On a stable prescribed standard of care (SoC) treatment regimen according to local guidelines and the specific requirements for each disease
* Systolic blood pressure ≤160 mmHg and diastolic blood pressure ≤90 mmHg at Screening. For participants aged ≥10 to <18 years, the average of 3 separate systolic and/or diastolic blood pressures <95th percentile for age, gender, and height

Diagnosis of IgAN, IgAVN, pMN, MCD, FSGS, or primary nephrotic syndrome

For patients enrolling in IgAN cohorts (eligibility varies by cohort):

* Age ≥ 10 years
* Biopsy proven IgAN or IgAVN,
* UPCR ≥ 0.5 g/g
* eGFR≥ 20 mL/min/1.73m2

For patients enrolling in pMN cohorts (eligibility varies by cohort):

* Age ≥ 18 years
* Biopsy-proven pMN
* Anti PLA2R antibodies ≥ 25 RU/mL
* UPCR ≥ 1.5 g/g
* At low risk for spontaneous remission (based on severity or duration of disease)

For patients enrolling in Nephrotic Syndrome cohorts (MCD, FSGS, or pediatric idiopathic nephrotic syndrome):

* Age ≥ 10 years
* eGFR≥30 mL/min/1.73m2
* Biopsy diagnosis of primary MCD or FSGS (adults) or challenging clinical course with steroids in children (frequenlty relapsing, steroid-dependent, or steroid-resistant)
* UPCR ≥ 1.0 g/g at Screening,
* Evidence of anti-nephrin antibodies

Key Exclusion Criteria

* Evidence of rapidly progressive glomerulonephritis (loss of ≥50% of eGFR) within 3 months prior to and at Screening)
* Active viral or bacterial infections
* Existing conditions or clinically significant laboratory abnormalities that may interfere with participation in this study
* Administration of live and live-attenuated vaccinations within 30 days prior to enrollment
* Known hypersensitivity to atacicept or any component of the formulated atacicept
* Additional criteria apply to each cohort/disease.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
AE profile and results of routine clinical and laboratory tests | Baseline until end of study: 52 + 26 Weeks
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), study drug discontinuation due to TEAEs
Percent reduction in urine protein to creatinine ratio (UPCR) | Baseline, Week 36
  Changes in proteinuria based on UPCR from 24 hour urine samples at baseline versus week 36

SECONDARY OUTCOMES:
Changes from baseline estimated glomerular filtration rate (eGFR). | Baseline, Week 36, Week 52
  Changes from baseline in estimated glomerular filtration rate (eGFR).
Change in disease-specific antibodies | Baseline through 52 Weeks
  IgAN: Percent change from baseline galactose-deficient IgA1 (GdIgA1) levels at 36 and 52 weeks.
  pMN: Percent change from baseline in anti-PLA2R antibody levels at 4, 8, 12, 36, and 52 weeks.
  MCD/FSGS: Percent change from baseline anti-nephrin antibody levels at 4, 8, 12, 36, and 52 weeks (exploratory).

CONTACTS AND LOCATIONS:
Overall Officials: Pam Winterberg, Study Director — Vera Therapeutics
Locations (1):
- Vera Therapeutics, Brisbane, California, United States